CLINICAL TRIAL: NCT00947739
Title: Phase I and Pharmacology Study of Camptothecin-20-O-Propionate Hydrate (CZ48) in Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Christus Stehlin Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST CZ48-01; NCI-2011-02688 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Advanced Solid Tumors; Lymphomas
Keywords: CZ; Stehlin; Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Cohort 1 (Experimental): 80 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48)PO, DAILY
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 2 (Experimental): 160 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, DAILY
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 3 (Experimental): 320 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, DAILY
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 4 (Experimental): 640 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, DAILY
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 5a (Experimental): 1280 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, DAILY
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 6 (Experimental): 2560 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 7 (Experimental): 18 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 8 (Experimental): 36 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 9 (Experimental): 72 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 10 (Experimental): 144 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 11 (Experimental): 288 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 12 (Experimental): 576 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 13 (Experimental): 750mg/m2 PO Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 14 (Experimental): 1000mg/m2 PO Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)
- Cohort 5b (Experimental): 1280 mg/m2 Camptothecin-20-O-Propionate Hydrate (CZ48) PO, TID
  Interventions: Drug: Camptothecin-20-O-Propionate Hydrate (CZ48)

INTERVENTIONS:
Drug: Camptothecin-20-O-Propionate Hydrate (CZ48) — CZ48 will be administered in successive cohorts of 1 patient per participating site until hints of toxicity (grade 2 or worse adverse events related to the drug) are observed. Then cohort of 3+3 patients will be treated. CZ48 will be administered orally daily for 3 weeks followed by a 1 week rest. (1 course = 4 weeks). No pre-medications will be administered. Patients will be asked to drink 2 liters of fluid daily to flush the bladder.
  Other Names: CZ48

SUMMARY:
This is a phase I and pharmacology study of Camptothecin-20-O-Propionate Hydrate (CZ48) in Patients with Solid Tumors or Lymphoma.

OBJECTIVES

Primary:

1. To describe the dose limiting toxicities and adverse event profile of Camptothecin-20-O-Propionate hydrate (CZ48) administered orally every day.
2. To determine Phase II recommended dose of Camptothecin-20-O-Propionate hydrate (CZ48) administered orally every day.

   Secondary:
3. To perform a pharmacokinetic study of orally administered CZ48 in the plasma.
4. To assess responses by RECIST criteria.
5. To follow patients for survival.

DETAILED DESCRIPTION:
CZ48 is an analog of the topoisomerase I inhibitor Camptothecin (CPT). CPT is an alkaloid extracted from the Chinese tree, Camptotheca acuminata. Only the S isomer (the natural form) is biologically active. The intact E lactone ring, which tends to be preserved in an acid environment, is essential for anti-tumor activity. Moreover, the open lactone ring moiety tends to promote toxicity [1-3]. In phase I and II trials conducted from 1970-1972 with the sodium salt of CPT (later shown to be largely inactive) toxicities included myelosuppression, diarrhea and cystitis [2, 3].

With the observation in 1984 that the mechanism of action of CPT was through topoisomerase I inhibition [1], renewed interest in the drug led to the development of a variety of analogs, some of which had higher potency than the parent drug. Some derivatives are water soluble such as CamptosarÂ® (irinotecan, CPTÂ¬-11) and HycamptinÂ® (topotecan), which are currently approved for use in the USA for colon and ovarian cancers, respectively. Studies have shown that substitutions at the C-9 and C- 10 positions enhance activity, and may confer water solubility. In general, analogs that are water-soluble have reduced anti-cancer activity in preclinical models.

The water-insoluble native camptothecin (CPT) caused diarrhea, which proved to be the dose limiting toxicity. Measurements demonstrated very little closed lactone ring CPT in the plasma of subjects receiving this compound [4]. This was later explained by the demonstration that CPT binds to human albumin, an action which promotes opening of the lactone ring [5]. Mouse albumin is much less efficient in this activity, hence explaining the greater antitumor activity observed in mice models.

In contrast to CPT, CZ48 incubated in vitro with human plasma and studied in vivo maintains a substantial closed lactone ring concentration in the plasma. It appears to act as a pro-drug. The removal of the side chain by endogenous esterases liberates the active drug, CPT. Malignant cells have a high esterase content and are rapidly transforming the pro-drug into the active parent drug. Preclinical studies suggest retention of anti-cancer activity and reduction in toxicity, probably because the pro-drug in the systemic circulation has no or little activity. Therefore, delivery of higher concentrations of closed lactone ring CPT analog inside the tumor cells should potentiate the anti-tumor activity. This study offers an opportunity to evaluate this hypothesis.

- OVERVIEW OF NONCLINICAL TESTING STRATEGY

All nonclinical pharmacology, pharmacokinetic, and toxicology studies described herein were conducted by or for The CHRISTUS Stehlin Foundation for Cancer Research. For studies conducted in accordance with GLP regulations, the location of records for inspection is/will be included in each study report. For nonGLP studies, study records are retained on file at:

The CHRISTUS Stehlin Foundation for Cancer Research 1315 St. Joseph Parkway, Suite #1818 Houston, TX 77002

Several experiments were conducted to examine the primary pharmacodynamics (i.e., efficacy and potency) of CZ48 against various tumor lines both in vitro and in vivo. In light of the intended Phase I patient population, the CZ48 safety pharmacology package was limited to in vitro and in vivo cardiovascular assessments. No secondary pharmacodynamic or pharmacodynamic drug interaction studies were conducted with CZ48.

Note: For all GLP studies the purity of the CZ48 as determined by HPLC validated methods is 98.9%. For these studies, the drug was formulated in a 0.5% medium density carboxymethyl cellulose aqueous suspension (CMC). For all non-GLP studies the drug (98% purity) was formulated as a suspension in cottonseed oil (except the non-GLP study performed by Covance which also used the CMC formulation).

Studies characterizing the pharmacokinetics and toxicokinetics of CZ48 and its active metabolite camptothecin after either single- or repeat-dose administration were conducted in mice and dogs. The repeat-dose studies were toxicokinetic evaluations conducted as part of the pivotal toxicology program using validated bioanalytical methods. No extensive distribution studies were conducted with CZ48; however, drug distribution into tumor, liver and kidney tissues of tumor-bearing mice was evaluated. Several in vitro and in vivo metabolism studies were conducted to examine the metabolic conversion of CZ48 to its active moiety, camptothecin. Excretion studies were limited to measurement of CZ48 in the feces of nude mice following single-dose administration. Pharmacokinetic drug interaction studies were not conducted with CZ48.

The CZ48 toxicology program consisted of exploratory (nonGLP) dose range-finding studies in the mouse and dog and definitive (GLP) toxicity and toxicokinetic studies in both species. Pivotal toxicology studies conducted with CZ48 employed the intended clinical route and schedule of administration. Additionally, two studies (nonGLP) were conducted in mice to assess the general tolerability of chronic high-dose CZ48 administration.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older, with incurable advanced solid tumors or lymphomas are eligible.
2. Patients must have a Zubrod performance status of 0-1.
3. Patients must sign an informed consent document.
4. Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 -along with an absence of a red blood cell transfusion in the two weeks prior to their participation in the trial.
5. Patients should have adequate hepatic function with a total bilirubin within normal range and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine within the upper limit of normal.
6. Patients may receive no other concurrent anticancer treatments such as chemotherapy, hormonotherapy (except for prostate cancer patients on LHRH agonists), immunotherapy, biological agents, investigational agents, or radiation therapy during this trial, and should be off these treatments for at least 2 weeks, or until they have completely recovered from the side effects of these treatments, whichever is longest, except for persistent grade 1 neuropathy in patients who received prior platinum or taxanes.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded from this study.
2. Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception (contraceptive pill, or IUD, or two mechanical barriers).
3. Patients with severe uncontrolled medical problems are not eligible for this trial.
4. Patients who have too much esterase activity in the blood, with a conversion rate yielding concentration of CPT > 20 ng/ml in vitro. Please see section 6.5 for sample collection, preparation and shipping. A validated analysis will be performed according to Sponsor SOP SFCR.PH.R.01.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To describe the dose limiting toxicities, adverse event profile, and Phase II recommended dose of Camptothecin-20-O-Propionate hydrate (CZ48). | 3 weeks

SECONDARY OUTCOMES:
To perform a pharmacokinetic study of orally administered CZ48 in the plasma. To assess responses by RECIST criteria and to follow patients for survival. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Monte Shaheen, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Texas Health Sciences Center, San Antonio, Texas

REFERENCES:
- See also: University of New Mexico Cancer Center — http://cancer.unm.edu
- See also: University of Texas Health Sciences Center — http://www.uth.edu/ctrc/